CLINICAL TRIAL: NCT06607393
Title: CARE Initiative Study: Real-world Emulation of the KEYNOTE-189 Comparative Effectiveness Trial of Pembrolizumab, Pemetrexed, and Chemotherapy vs. Placebo, Pemetrexed, and Chemotherapy for the First-line Treatment of Metastatic Non-small Cell Lung Cancer
Brief Title: CARE Initiative: Real-world Emulation of the KEYNOTE-189 Trial [DS3]
Status: Completed | Type: Observational
Sponsor: Aetion, Inc. (Other)
Collaborators: AbbVie (Industry); Amgen (Industry); AstraZeneca (Industry); Bayer (Industry); Gilead Sciences (Industry); Janssen, LP (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: DS3-KN189
Record Dates: First submitted 2024-09-03; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Nonsmall Cell Lung Cancer
Keywords: real-world evidence; real-world data; oncology; pharmacoepidemiology; comparative effectiveness research; trial emulation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — pembrolizumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed: Patients initiating pemetrexed, cisplatin or carboplatin, and pembrolizumab as first-line treatment for metastatic NSCLC
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Comparator: Patients initiating pemetrexed and cisplatin or carboplatin as first-line treatment for metastatic NSCLC
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab
  Groups: Exposed
Drug: Pemetrexed
Drug: Cisplatin
Drug: Carboplatin

SUMMARY:
The goal of this non-interventional study is to emulate the KEYNOTE-189 randomized controlled trial of pembrolizumab for the treatment of metastatic non-small cell lung cancer using real-world, electronic health record data. The main questions this study aims to answer are:

1. Do patients with metastatic non-small cell lung cancer (NSCLC) treated with pemetrexed, cisplatin/carboplatin, and pembrolizumab have improved real-world overall survival (rwOS) and real-world progression-free survival (rwPFS) compared with patients treated with pemetrexed and cisplatin/carboplatin alone?
2. How do the results of this non-interventional study compare to those of the KEYNOTE-189 randomized controlled trial?

DETAILED DESCRIPTION:
The Coalition to Advance Real-World Evidence through Randomized Controlled Trial Emulation (CARE) Initiative is a program designed to build an empirical evidence base for the use of real-world data (RWD) in clinical and regulatory decision-making. Using randomized controlled trials (RCTs) as a benchmark for causal effect estimates, a series of RCT emulations will be conducted across varying trials, real world data sources, and study design elements to better understand under what conditions non-interventional studies, using data generated during routine clinical care, can provide reliable conclusions about drug effectiveness.

In this study, real-world electronic health record (EHR) data will be used to emulate the KEYNOTE-189 efficacy trial of pembrolizumab as first-line therapy in patients with metastatic non-small cell lung cancer (NSCLC) without epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) sensitizing mutations. Similarly to the KEYNOTE-189 trial, this study will compare real-world overall survival (rwOS) and real-world progression-free survival (rwPFS) between patients who initiate pemetrexed, platinum-based chemotherapy, and pembrolizumab, and patients who initiate pemetrexed and platinum-based chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) diagnosis
* Histology not indicative of squamous cell carcinoma
* Metastatic disease
* Epidermal growth factor receptor (EGFR) and Anaplastic lymphoma kinase (ALK)-negative or Kirsten rat sarcoma viral oncogene homolog (KRAS)-positive
* No prior systemic treatment for metastatic NSCLC
* No record of adjuvant or neoadjuvant therapy in the 12 months before metastatic diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or missing or Karnofsky performance status >=70 or missing
* No lab results indicating inadequate organ function, as defined in the KEYNOTE-189 RCT protocol

Exclusion Criteria:

* Histology indicative of squamous cell carcinoma or small cell elements
* Prior systemic treatment for metastatic NSCLC
* Prior antineoplastic biological therapy
* History of major cancer-related surgery in the 3 weeks before study drug initiation
* Radiation therapy to the lung >30 Gy in the 6 months before study drug initiation
* Prior diagnosis of clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction
* Diagnosis of a second primary malignant neoplasm
* Diagnosis of brain, central nervous system, and/or spinal cord metastases
* Diagnosis of autoimmune disease and treatment with corticosteroids or immunosuppressive drugs after diagnosis and within the 2 years prior to study drug initiation
* Treatment with a non-topical systemic steroid in each of the 6 months prior to study drug initiation
* Prior treatment with pembrolizumab or any other anti-PD-1, PD-L1, PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Treatment with non-topical antibiotics, antifungals, or antivirals within 2 weeks after an infection diagnosis in the month prior to study drug initiation
* Diagnosis of human immunodeficiency virus infection
* Diagnosis of acute hepatitis B or C
* Diagnosis of ascites or plural effusion in the 3 months prior to study drug initiation
* Prior diagnosis of interstitial lung disease or diagnosis of pneumonitis and record of treatment with glucocorticoids within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified in the electronic health record data source with metastatic EGFR/ALK-negative non-small cell lung cancer initiating treatment with the study drugs (pemetrexed, cisplatin/carboplatin, pembrolizumab)
Sampling Method: Non-Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Real-world overall survival (rwOS) | From study treatment initiation until the date of death from any cause or censoring, whichever came first, assessed up to 20.4 months.
  Time from study treatment initiation to death
Real-world progression-free survival (rwPFS) | From study treatment initiation until the date of disease progression, death from any cause or censoring, whichever came first, assessed up to 20.4 months.
  Time from study treatment initiation to disease progression or death

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT06607393/Prot_SAP_000.pdf